CLINICAL TRIAL: NCT04680611
Title: The Biopsychosocial Impact of Mepolizumab in Severe Eosinophilic Asthma on Quantitative and Qualitative Emotional and Affective Outcomes in Patients and Partners
Brief Title: Severe Asthma, MepolizumaB and Affect: SAMBA Study
Acronym: SAMBA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); University of Derby (Other)
Responsible Party: Sponsor
Other Study IDs: RHM MED1740
Record Dates: First submitted 2020-12-08; First posted 2020-12-23 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Severe Eosinophilic Asthma; Psychological Distress; Anxiety; Depression; Psychological Stress; Psychological Adjustment; Psychological Disorder; Psychosocial Problem; Psychosocial Stressor; Psychological; Emotions; Emotional Disorder; Emotional Dysfunction; Emotional Distress; Adjustment; Adjustment, Emotional; Coping Behavior
MeSH Terms: conditions — Pulmonary Eosinophilia; Anxiety Disorders; Depression; Stress, Psychological; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — inflammatory panel, chemokines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with severe eosinophilic asthma Phase 1: Patients with severe eosinophilic asthma on Nucala(R) treatment
  Interventions: Other: no study intervention. Patients receive standard clinical care
- Patients with severe eosinophilic asthma Phase 2: Patients with severe eosinophilic asthma to start Nucala(R) treatment
  Interventions: Other: no study intervention. Patients receive standard clinical care
- Partners of patients with severe eosinophilic asthma Phase 2: Partners of patients with severe eosinophilic asthma to start Nucala(R) treatment
- Phase 3: Patients with severe eosinophilic asthma from Phase 2: A sub-group of patients who participate in Phase 2
  Interventions: Other: no study intervention. Patients receive standard clinical care
- Phase 3: Partners of patients in Phase 3: Partners of the sub-group of patients who participate in Phase 3

INTERVENTIONS:
Other: no study intervention. Patients receive standard clinical care — no intervention. observational study
  Other Names: no intervention. observational study
  Groups: Patients with severe eosinophilic asthma Phase 1; Patients with severe eosinophilic asthma Phase 2; Phase 3: Patients with severe eosinophilic asthma from Phase 2

SUMMARY:
This is a real-life pragmatic non-randomised study to explore the impact of mepolizumab on the emotional and affective outcomes of patients with severe eosinophilic asthma and their partners. It will be conducted in two quantitative stages (Phases 1 and 2) with an additional third qualitative component (Phase 3).

DETAILED DESCRIPTION:
This longitudinal observational study will investigate the relationship between patients' asthma control and emotional states and quality of life in patients and their partners where patients have severe eosinophilic asthma. The study will consist of three phases.

Phase 1 In order to extend our pilot study findings and help inform the second stage, investigators will gather Geneva Emotional Wheel (GEW) data from 30 patients currently treated and benefitting from mepolizumab (Nucala®). This data will be compared to the GEW data investigators have already gathered from patients with severe asthma not receiving treatment with mepolizumab (Nucala®). This will provide timely data to support a publication on the GEW findings in severe asthma and allow the description of the impact of mepolizumab (Nucala®). In addition, it will help provide power calculations for a prospective study. Parallel assessment of quality of life (SGRQ and SAQ) and anxiety and depression (HADS) will be made to evaluate the relationship between GEW, SGRQ, SAQ and HADS scores.

Phase 2 In the second stage, investigators will conduct a prospective study of 45 patients newly prescribed mepolizumab (Nucala®) and their partners measuring participants' emotional composition before and 6 and 12 months after starting treatment. The choice of 60 has been based on likely power requirements but was adjusted to 45 based in Phase 1 results. Investigators will also compare the outcomes from the GEW with other standard outcome measures (HADS, ACQ, SGRQ, SAQ, BIPQ), to establish relationship between changes in these measures and changes in GEW scores, to evaluate the utility of the GEW. This will help determine if the GEW reflects changes in asthma control or whether it is reflecting improvements that the current established instruments do not recognise and allow us to quantify the magnitude of that effect. As these patients will receive mepolizumab as part of their clinical care for a year, whilst assessment of clinical efficacy is being established, investigators will gather data on oral steroid dependent exacerbations (severe exacerbations) during this year and relate to their historic exacerbation history in the year before. Evaluation will be made as to whether the 6-month improvement in GEW scores predicts impact of mepolizumab on exacerbation reduction over the first year of administration. In addition, improvements in the GEW will be explored in relationship to systemic inflammatory impact, with measures of blood eosinophils and serum inflammatory biomarkers (Olink inflammatory panel) at baseline, 6 months and 1 year.

Phase 3 Finally, in addition, investigators will conduct qualitative research in the form of semi-structured interviews with a sub-set of couples (20 couples or less if no new information emerges from the interviews) to gain a more detailed insight and identify common key aspects in their subjective experiences, quality of life and emotional processes before starting treatment and after being on treatment with mepolizumab for 6 months.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Age 18 or over
* Having a diagnosis of severe eosinophilic asthma
* Currently on mepolizumab (Nucala®) treatment
* At least basic command of English
* Giving written informed consent

Phase 2 Patient eligibility Inclusion criteria

* Age 18 or over
* Having a diagnosis of severe eosinophilic asthma
* Scheduled to start mepolizumab (Nucala®) treatment
* At least basic command of English (for sub-study: conversational level of English that does not require a translator)
* Giving written informed consent
* Co-habiting with an intimate partner who is willing to participate in the study

Exclusion criteria

* Participated in Phase 1
* Currently on mepolizumab (Nucala®) treatment
* Major psychiatric disorder currently under treatment
* History of any major psychiatric disorder in the last 5 years, excluding depressive and anxiety disorders that can be included if treatment or change of treatment (including change in dose of medication) has not started within the last 6 months
* Any diagnosed severe comorbid chronic condition that, in the opinion of the patient's asthma physician, might impact on the patient's or partner's affective state (e.g. cancer, diabetes, heart failure, chronic liver disease, chronic kidney disease, autoimmune or neuro-degenerative disease).
* Partners only: diagnosis of severe eosinophilic asthma
* Death of spouse, main informal carer or first-degree family member within the last 3 months
* Current oral corticosteroid maintenance treatment

Partner eligibility Inclusion criteria

* Age 18 or over
* At least basic command of English (for sub-study: conversational level of English that does not require a translator)
* Giving written informed consent
* Partners: Co-habiting with an intimate partner who has severe eosinophilic asthma and is willing to participate in the study

Exclusion criteria

* Participated in Phase 1
* Major psychiatric disorder currently under treatment
* Participant self-reported history of any major psychiatric disorder in the last 5 years, excluding depressive and anxiety disorders that can be included if treatment or change of treatment (including change in dose of medication) has not started within the last 6 months.
* Participant self-reported any diagnosed severe comorbid chronic condition that, in the opinion of the patient's asthma physician, might impact on the patient's or partner's affective state (e.g. cancer, diabetes, heart failure, chronic liver disease, chronic kidney disease, autoimmune or neuro-degenerative disease).
* Diagnosis of severe eosinophilic asthma
* Death of spouse, main informal carer or first-degree family member within the last 3 months
* Current oral corticosteroid maintenance treatment

Phase 3:

Phase 3 is a qualitative study on a sample of couples from Phase 2 therefore the same exclusion criteria will apply as in Phase 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe eosinophilic asthma on mepolizumab treatment (Phase 1) Patients with sereve eosinophilic asthma who are to start mepolizumab treatment and their partners ( Phase 2 and 3)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in emotional composition (using the Geneva Emotions Wheel) | Phase 1: on enrolment. Phase 2: change to one year after start of treatment
  A 20-item self-report questionnaire identifying 20 discrete emotions with positive or negative valence. The intensity of each emotion can be marked on a 6-point Likert-type scale. Lower scores indicate lower intensity of emotions, higher scores indicate higher intensity of emotions. Respondents can add free text. Can be used a a variety of applications. The emotion labels used in the study have been modified with input from representatives of the target study population to ensure complete relevance to the study..

SECONDARY OUTCOMES:
change in affective state (using the Hospital Anxiety and Depression Scale) | Phase 1: on enrolment. Phase 2: change from baseline to 1 year after start of treatment
  Clinical diagnostic self-report questionnaire to assess psychological distress. Consists of anxiety and depression sub-scales. It consists of seven questions for anxiety and seven questions for depression that are in mixed order in the questionnaire. Each question has four possible answers scored from 0-3. There are separate sub-scale scores for anxiety and depression each with cut-off scores 0-7: normal, 8-10: borderline abnormal and 11-21: abnormal. The HADS is a self-report tool and takes 2-5minutes to complete.
change in self-reported asthma symptom control (using the Asthma Control Questionnaire) | Phase 1: on enrolment. Phase 2: change from baseline to 1 year after start of treatment
  6-item clinical questionnaire to establish self-assessed asthma control (questions 1-6) and lung function measured by healthcare professional (item 7). 6 of the questions are patients self-report about their asthma during the previous week regarding symptoms and bronchodilator use. Responses are given on a 7-point scale (0=no impairment, 6= maximum impairment). The ACQ score is the mean of all the questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). In general, patients with a score below 1.0 have adequately controlled asthma and above 1.0 their asthma is not controlled. Patients with a score between 0.75 and 1.25 have borderline of adequate control. The smallest clinically important change is 0.5.
change in functioning and quality of life (using the St Georges Respiratory Questionnaire) | Phase 1: on enrolment Phase 2: change from baseline to 1 year after start of treatment
  Clinical questionnaire to assess disease impact on quality of life. QThe questionnaire has two parts. Part 1 (Questions 1 to 8) covers the patients' recollection of their symptoms over the preceding period (range 1 month to 1 year). Part 2 (Questions 9 to 16) is related to the patients' current state. The Activity score covers functioning related to patients' daily physical activity. The Impacts score relates to psychosocial functioning. Although this component relates partly to physical symptoms, it also correlates quite strongly with exercise performance, breathlessness and disturbances of mood (anxiety and depression), therefore it is the broadest component of the questionnaire, covering the whole range of disturbances that respiratory patients experience in their lives. Scoring is weighted, gihres scores indicate worse outcomes.
change in asthma-related quality of life (using the Severe Asthma Questionnaire) | Phase 1: on enrolment Phase 2: change from baseline to 1 year after start of treatment
  Questionnaire assessing the impact of severe asthma and the effects of treatment on patient's self-reported health-related quality of life. The questionnaire produces two scores: the SAQ score is the aggregation of 16 different QoL domains and the SAQ-global score is the figure given on a 100-point scale. Higher scroes indicate higher adverese impact on the responder's life.The scale takes between 3 to 6 minutes to complete, but completion time reduces on subsequent occasions.
change in illness perception (using the Brief Illness Perception Questionnaire) | Phase 2: change from basline to 1 year after start of treatment
  Questionnaire assessing the beliefs individuals have about the cause, controllability and impact on them of the illness. Comprises 9 questions. 8 questions use a Likert scale response. Question 9 can be answered by free text about the perceived cause of illness.

OTHER OUTCOMES:
change in Inflammatory panel and chemokines | Phase 2 only: change from baseline to 1 year after start of treatment
  Olink inflammatory panel and particular chemokines that are comprehensively listed at https://www.olink.com/content/uploads/2019/04/Olink-Inflammation-Validation-Data-v3.0.pdf) will be used to measure markers of systemic inflammation and assess links between affective states and systemic inflammation. In addition, Serum CCl17 and CCL26 will be measured by ELISA as these biomarkers do not feature in the Olink inflammatory panel.
lived experiences and psychological processes (using Semi-structured interviews) | Phase 2 only: change from baseline to 1 year after start of treatment
  Interviews to explore participants' quality of life

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Department of Respiratory Medicine, Aberdeen Royal Infirmary, Aberdeen, Grampian
  - Judit Varkonyi-Sepp, Southampton, Hampshire
  - Hull University Teaching Hospitals NHS Trust, Hull, Yorkshire
  - Pinderfields Hospital, Wakefield, Yorkshire
  - Glasgow Gartnavel General Hospital, Glasgow
  - Portsmouth Hospitals NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No
Only anonymised and aggregate data will be shared